CLINICAL TRIAL: NCT02472249
Title: Hepatic Arterial Blood Flow Modulation in Patients With Hepatocellular Carcinoma: Influence of Intra-arterial Norepinephrine Assessed With CT Perfusion
Brief Title: Pharmacological Manipulation of Intrahepatic Arterial Blood Flow in HCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-8122-C
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: TACE; CT perfusion; Liver blood flow
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cytidine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Norepinephrine intra-arteriel/hepatic (Experimental): This is the only arm of this study. These patients will receive 24 micrograms of norepinephrine in the hepatic artery with subsequent CT perfusion imaging to evaluate liver blood flow.
  Interventions: Radiation: CT perfusion; Drug: Norepinephrine intra-arteriel/hepatic

INTERVENTIONS:
Radiation: CT perfusion — Two dynamic CT perfusion acquisitions of the whole liver will be performed with a 320-detectors CT, prior and after to the norepinephrine injection.
Drug: Norepinephrine intra-arteriel/hepatic — A small dose (24 ug) of norepinephrine will be injected in the hepatic artery over 10 seconds. The half-life of the drug is 90 seconds..

SUMMARY:
Dr Rajan is investigating a new method to improve local treatment of liver cancer. There is evidence that a drug, norepinephrine (NE), has the ability to shrink down normal liver blood vessels, but leave tumor vessels wide open. In patients with primary liver cancer, NE will be injected directly in the artery that nourishes the liver and the tumor. Real time blood flow will be measured using an advanced CT scanner to demonstrate the NE effect on blood vessels. If Dr Rajan's hypothesis is confirmed, this drug has great potential to benefit patients during local delivery of chemotherapy in the liver artery, diverting it away from normal liver and towards the tumor, resulting in less complications and improved tumor kill.

DETAILED DESCRIPTION:
This study aims to evaluate the blood flow modifications in liver following injection of norepinephrine in the hepatic artery. These blood flow variations have never been dynamically evaluated before. If indeed blood flow modulation in liver is favorable, the use of norepinephrine prior to localized chemotherapy has great potential to enhance treatment and diminish side effects. Patients with hepatocellular carcinoma, a primary liver cancer, will be selected for this study. Included patients will have a trans-arterial chemoembolization (TACE) procedure scheduled as treatment for their cancer. During their procedure, they will be brought to an advanced CT-scanner. CT perfusion imaging will be performed prior, and after the injection of the study drug in the liver artery. Patient's treatment will then be completed. Perfusion color maps will illustrate blood flow. Perfusion values will be correlated to see how the drug modulates blood flow in tumor and in normal liver.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven HCC< or confident diagnosis of HCC on multi-phasic CT or MRI
* Selection criteria for chemoembolization must be met, including adequate coagulation profile and serum creatinine, patent portal vein, no severe contrast allergy, cirrhosis Child A or B.
* 5 or less untreated nodular hepatic tumors within the lobe to undergo chemoembolization. Larger nodule must be equal or over 3 cm.
* Patient must be able to provide written, informed consent.

Exclusion Criteria:

* Symptoms or history of ischemic cardiac disease or arrhythmia
* Uncontrolled hypertension
* Pregnancy or desire to get pregnant
* Severe COPD, FEVS lower than 30%
* Prior documented hypersensitivity to norepinephrine
* Patients receiving MAO inhibitors, or anti-depressants of the triptyline or imipramine types

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Liver blood flow | 1 minute following injection
  Liver blood flow as measured with CT perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Dheeraj Rajan, MD FRCPC, Principal Investigator — University Health Network/Mount Sinai Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada